CLINICAL TRIAL: NCT02048371
Title: SARC024: A Blanket Protocol to Study Oral Regorafenib in Patients With Selected Sarcoma Subtypes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SARC024
Record Dates: First submitted 2014-01-10; First posted 2014-01-29 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Liposarcoma; Osteogenic Sarcoma; Ewing/Ewing-like Sarcoma; Rhabdomyosarcoma; Mesenchymal Chondrosarcoma
MeSH Terms: conditions — Liposarcoma; Osteosarcoma; Rhabdomyosarcoma; Chondrosarcoma, Mesenchymal | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort A: Liposarcoma (Active Comparator): Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Interventions: Drug: Regorafenib
- Cohort A: Liposarcoma, Placebo (Placebo Comparator): 21 days on and 7 days off
  Placebo
  Interventions: Drug: Placebo
- Cohort B: Osteosarcoma (Active Comparator): Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Interventions: Drug: Regorafenib
- Cohort B: Osteosarcoma, placebo (Placebo Comparator): 21 days on and 7 days off
  Placebo
  Interventions: Drug: Placebo
- Cohort C: Ewing sarcoma (Active Comparator): Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Interventions: Drug: Regorafenib
- Cohort D: Rhabdomyosarcoma (Active Comparator): Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Interventions: Drug: Regorafenib
- Cohort E: Mesenchymal Chondrosarcoma (Active Comparator): Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Arms: Cohort A: Liposarcoma; Cohort B: Osteosarcoma; Cohort C: Ewing sarcoma; Cohort D: Rhabdomyosarcoma; Cohort E: Mesenchymal Chondrosarcoma
Drug: Placebo — 21 days on and 7 days off
  Arms: Cohort A: Liposarcoma, Placebo; Cohort B: Osteosarcoma, placebo

SUMMARY:
Although regorafenib was approved for use in patients who had progressive GIST despite imatinib and/or sunitinib on the basis of phase II and phase III data, it has not been examined in a systematic fashion in patients with other forms of sarcoma.

Given the activity of sorafenib, sunitinib and pazopanib in soft tissue sarcomas, and evidence of activity of sorafenib in osteogenic sarcoma and possibly Ewing/Ewing-like sarcoma, there is precedent to examine SMOKIs (small molecule oral kinase inhibitors) such as regorafenib in sarcomas other than GIST. It is also recognized that SMOKIs (small molecule oral kinase inhibitors)such as regorafenib, sorafenib, pazopanib, and sunitinib have overlapping panels of kinases that are inhibited simultaneously. While not equivalent, most of these SMOKIs (small molecule oral kinase inhibitors) block vascular endothelial growth factor and platelet derived growth factors receptors (VEGFRs and PDGFRs), speaking to a common mechanism of action of several of these agents.

DETAILED DESCRIPTION:
Although regorafenib was approved for use in patients who had progressive GIST despite imatinib and/or sunitinib on the basis of phase II and phase III data, it has not been examined in a systematic fashion in patients with other forms of sarcoma.

Given the activity of sorafenib, sunitinib and pazopanib in soft tissue sarcomas, and evidence of activity of sorafenib in osteogenic sarcoma and possibly Ewing/Ewing-like sarcoma, there is precedent to examine SMOKIs (small molecule oral kinase inhibitors) such as regorafenib in sarcomas other than GIST. It is also recognized that SMOKIs (small molecule oral kinase inhibitors)such as regorafenib, sorafenib, pazopanib, and sunitinib have overlapping panels of kinases that are inhibited simultaneously. While not equivalent, most of these SMOKIs (small molecule oral kinase inhibitors) block vascular endothelial growth factor and platelet derived growth factors receptors (VEGFRs and PDGFRs), speaking to a common mechanism of action of several of these agents

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 10 year for Liposarcoma, Osteosarcoma, Ewing sarcoma and Mesenchymal Chondrosarcoma; Age ≥ 5 years for Rhabdomyosarcoma cohorts
* Weight ≥ 15 kg (33 lb)
* Patients must have histologically or cytologically confirmed advanced/metastatic liposarcoma, osteogenic sarcoma, Ewing/Ewing-like sarcoma of soft tissue or bone, fusion-positive alveolar rhabdomyosarcoma or embryonal rhabdomyosarcoma/fusion-negative alveolar rhabdomyosarcoma , or mesenchymal chondrosarcoma
* WHO Performance Status 0, 1 or 2. A maximum of 1/3 of patients in cohorts A & B may be WHO performance status 2
* At least one prior line of systemic therapy for the sarcoma diagnosis (neoadjuvant, adjuvant or metastatic disease)
* All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v 4.0 Grade 1 or less (except alopecia) at the time of signing the Informed Consent Form (ICF)
* Subject must be able to swallow and retain oral medication
* At least one site of measurable disease on x-ray/CT/MRI scan as defined by RECIST 1.1
* Adequate organ function within 14 days of registration
* Written, voluntary informed consent
* Fertile men and women of childbearing potential must agree to use an effective method of birth control from Day 1 of study and for 3 months after last study drug administration in both sexes, as assessed by the investigator. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test less than or equal to seven days prior to Day 1 of study. The definition of adequate contraception will be based on the judgement of the investigator.
* Evidence of progression of disease as defined by RECIST 1.1 (i.e. new disease sites or 20% growth of index lesions) within 6 months of registration
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of CNS (central nervous system) metastatic disease and are without evidence of clinical progression for at least 12 weeks after therapy

Exclusion Criteria:

* Patients with documentation of well differentiated liposarcoma only (of the well differentiated/dedifferentiated liposarcoma family) are specifically excluded, owing to its characteristically slow growth. If high grade areas are suspected (dedifferentiation), but not proved by pathology analysis (e.g. after primary resection of a well-differentiated liposarcoma), a biopsy must be performed to demonstrate the high-grade dedifferentiated disease
* Prior systemic therapy with a small molecule oral kinase inhibitor, including but not limited to: pazopanib, sunitinib, sorafenib, everolimus, sirolimus, vemurafenib, dasatinib and trametinib
* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study. Patients who progress on placebo are specifically allowed to enroll on the treatment arm of the study if they meet all other entry criteria
* Concurrent, clinically significant, active malignancies within 12 months of study enrollment
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* Major surgery within 28 days prior to study registration or those patients who have not recovered adequately from prior surgery
* Patients who have received wide field radiotherapy ≤ 28 days (defined as > 50% of volume of pelvis bones or equivalent) or limited field radiation for palliation < 14 days prior to study registration or those patients who have not recovered adequately from side effects of such therapy
* Patients who have received prior systemic therapy < 14 days prior to study registration or have not recovered adequately from toxicities to CTCAE v. 4.03 grade 1 or less; prior investigational therapy may not have been given < 5 half-lives of last dose of treatment, or < 14 days, whichever is greater
* Patients who have had prior autologous, or allogeneic bone marrow transplant
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v 4.0] on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease including: Congestive heart failure-New York Heart Association (NYHA) > class II, Active coronary artery disease, Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, Unstable angina (anginal symptoms at rest), new onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization
* Evidence or history of bleeding diathesis
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to study registration
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection > Grade 2 NCI-CTCAE v 4.03
* Presence of a non-healing wound, non-healing ulcer, or benign bone fracture (patients with stress insufficiency fractures e.g. from osteoporosis or pathological fracture from tumor are eligible for study)
* Patients with seizure disorder requiring medication
* Proteinuria > 100 mg/dl on urine analysis
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.03 Grade 2 dyspnea)
* History of organ allograft (including corneal transplant).
* Known or suspected allergy or hypersensitivity to regorafenib, or excipients of the formulations given during the course of this trial
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Inability to comply with protocol required procedures
* Use of any herbal remedy (e.g. St. John wort [Hypericum perforatum])

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (18):
- United States (18):
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Stanford University, Stanford, California
  - Mayo Clinic - Florida, Jacksonville, Florida
  - H. Lee Moffitt, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Dana Farber/Partners Cancer Care, Boston, Massachusetts
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Riedel RF, Ballman KV, Lu Y, Attia S, Loggers ET, Ganjoo KN, Livingston MB, Chow W, Wright J, Ward JH, Rushing D, Okuno SH, Reed DR, Liebner DA, Keedy VL, Mascarenhas L, Davis LE, Ryan C, Reinke DK, Maki RG. A Randomized, Double-Blind, Placebo-Controlled, Phase II Study of Regorafenib Versus Placebo in Advanced/Metastatic, Treatment-Refractory Liposarcoma: Results from the SARC024 Study. Oncologist. 2020 Nov;25(11):e1655-e1662. doi: 10.1634/theoncologist.2020-0679. Epub 2020 Aug 20. PMID 32701199
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903
- [Derived] Davis LE, Bolejack V, Ryan CW, Ganjoo KN, Loggers ET, Chawla S, Agulnik M, Livingston MB, Reed D, Keedy V, Rushing D, Okuno S, Reinke DK, Riedel RF, Attia S, Mascarenhas L, Maki RG. Randomized Double-Blind Phase II Study of Regorafenib in Patients With Metastatic Osteosarcoma. J Clin Oncol. 2019 Jun 1;37(16):1424-1431. doi: 10.1200/JCO.18.02374. Epub 2019 Apr 23. PMID 31013172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrollment ended early due to slow enrollment.
Groups:
- Cohort A: Liposarcoma; Cohort B: Osteosarcoma; Cohort C: Ewing Sarcoma; Cohort D: Rhabdomyosarcoma; Cohort E: Mesenchymal Chondrosarcoma: Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Regorafenib: Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
- Cohort A: Liposarcoma, Placebo; Cohort B: Osteosarcoma, Placebo: 21 days on and 7 days off
  Placebo
  Placebo: 21 days on and 7 days off
- Cohort A: Liposarcoma Crossover: Those patients who started on placebo and crossed over to active drug. Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Regorafenib: Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
- Cohort B: Osteosarcoma Crossover: Patients who started on placebo and crossed over to active drug.
  Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Regorafenib: Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
Period: Overall Study
Arm/Group | Cohort A: Liposarcoma | Cohort A: Liposarcoma, Placebo | Cohort A: Liposarcoma Crossover | Cohort B: Osteosarcoma | Cohort B: Osteosarcoma, Placebo | Cohort B: Osteosarcoma Crossover | Cohort C: Ewing Sarcoma | Cohort D: Rhabdomyosarcoma | Cohort E: Mesenchymal Chondrosarcoma
Started | 24 | 9 | 15 | 22 | 9 | 11 | 30 | 10 | 1
Completed | 17 | 1 | 9 | 11 | 3 | 8 | 22 | 6 | 1
Not Completed | 7 | 8 | 6 | 11 | 6 | 3 | 8 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Liposarcoma | Cohort A: Liposarcoma, Placebo | Cohort B: Osteosarcoma | Cohort B: Osteosarcoma, Placebo | Cohort C: Ewing Sarcoma | Cohort D: Rhabdomyosarcoma | Cohort E: Mesenchymal Chondrosarcoma | Total
Number analyzed (Participants) | 24 | 24 | 22 | 20 | 30 | 10 | 1 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
  Between 18 and 65 years | 17 | 12 | 21 | 16 | 29 | 6 | 1 | 102
  >=65 years | 7 | 12 | 1 | 4 | 1 | 0 | 0 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 16 | 6 | 10 | 5 | 0 | 57
  Male | 10 | 18 | 6 | 14 | 20 | 5 | 1 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 4 | 2 | 1 | 2 | 0 | 10
  Not Hispanic or Latino | 23 | 22 | 17 | 17 | 28 | 6 | 1 | 114
  Unknown or Not Reported | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 0 | 3 | 2 | 3 | 2 | 1 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 5 | 1 | 5 | 0 | 0 | 0 | 0 | 11
  White | 16 | 20 | 12 | 15 | 27 | 8 | 1 | 99
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS). Cohort A and Cohort B
Description: The progression-free survival is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. Cohort A (liposarcoma) and Cohort B (osteosarcoma). PFS will be evaluated according to RECIST (Response Evaluation Criteria In Solid Tumors) 1.1, where a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Liposarcoma | Cohort A: Liposarcoma, Placebo | Cohort B: Osteosarcoma | Cohort B: Osteosarcoma, Placebo
Number analyzed (Participants) | 24 | 24 | 22 | 20
months | 1.87 [0.92 to 3.67] | 2.07 [1.64 to 3.44] | 3.6 [2.0 to 7.6] | 1.7 [1.2 to 1.8]

2. Primary Outcome: Progression-free Survival (PFS). Cohort C, Cohort D, and Cohort E
Description: The progression-free survival is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. Cohort C (Ewing/Ewing-like sarcoma). PFS will be evaluated according to RECIST (Response Evaluation Criteria In Solid Tumors) 1.1.
Time Frame: up to 16 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort C: Ewing Sarcoma | Cohort D: Rhabdomyosarcoma | Cohort E: Mesenchymal Chondrosarcoma
Number analyzed (Participants) | 30 | 10 | 1
months | 3.4 [1.7 to 3.7] | 1.82 [1.58 to NA] — The upper limit of the CI is below the level of detection. | NA [NA to NA] — There is only one participant, so statistics cannot be calculated.

3. Secondary Outcome: The Number of Participants With Reported CTCAE (Common Terminology Criteria for Adverse Events) Version 4.03 Adverse Events. All Cohorts.
Description: Common Toxicity Criteria, also referred to as the Common Terminology Criteria for Adverse Events (CTCAE), is a standardized classification of side effects used in assessing drugs for cancer therapy. Cohorts A, B, C, and D.
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Liposarcoma | Cohort A: Liposarcoma, Placebo | Cohort B: Osteosarcoma | Cohort B: Osteosarcoma, Placebo | Cohort C: Ewing Sarcoma | Cohort D: Rhabdomyosarcoma | Cohort E: Mesenchymal Chondrosarcoma
Number analyzed (Participants) | 24 | 24 | 22 | 20 | 30 | 10 | 1
Participants | 12 | 15 | 6 | 9 | 6 | 2 | 0

4. Secondary Outcome: Overall Response Rate (ORR). All Cohorts.
Description: The overall response rate (ORR) is the percentage of patients whose cancer shrinks or disappears after treatment. ORR will be evaluated according to RECIST (Response Evaluation Criteria In Solid Tumors) 1.1
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Liposarcoma | Cohort A: Liposarcoma, Placebo | Cohort B: Osteosarcoma | Cohort B: Osteosarcoma, Placebo | Cohort C: Ewing Sarcoma | Cohort D: Rhabdomyosarcoma | Cohort E: Mesenchymal Chondrosarcoma
Number analyzed (Participants) | 24 | 24 | 22 | 20 | 30 | 10 | 1
Participants | 0 | 1 | 3 | 0 | 3 | 0 | 0

5. Secondary Outcome: Progression-free Survival (PFS), Cohorts A and B, After Crossover.
Description: The progression-free survival is the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Time Frame: up to 3 years
Population: Participants who started on placebo in Cohorts A and B, then crossed over to active drug after progression.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort A: Liposarcoma Crossover; Cohort B: Osteosarcoma Crossover: Participants who started on placebo and crossed over to active drug.
  Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Regorafenib: Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
Arm/Group | Cohort A: Liposarcoma Crossover | Cohort B: Osteosarcoma Crossover
Number analyzed (Participants) | 15 | 11
months | 1.68 [0.92 to 5.59] | 5.78 [3.55 to NA] — The upper limit of the CI is below the level of detection.

6. Secondary Outcome: Response Rate (RR), Cohorts A and B, After Crossover.
Description: The response rate (RR) is the percentage of patients whose cancer shrinks or disappears after treatment.
Time Frame: up to 3 years
Population: Participants who started on placebo then crossed over to active drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: Liposarcoma Crossover; Cohort B: Osteosarcoma Crossover: Participants who crossed over to active drug after placebo. Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Regorafenib: Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
Arm/Group | Cohort A: Liposarcoma Crossover | Cohort B: Osteosarcoma Crossover
Number analyzed (Participants) | 15 | 11
Participants | 0 | 0

7. Secondary Outcome: Time to Tumor Progression (TTP), Cohorts A and B, After Crossover.
Description: Time to tumor progression (TTP) is the length of time from the date of diagnosis or the start of treatment for a disease until the disease starts to get worse or spread to other parts of the body.
Time Frame: up to 3 years
Population: Participants who crossed over to active drug after placebo.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Liposarcoma Crossover | Cohort B: Osteosarcoma Crossover
Number analyzed (Participants) | 15 | 11
months | 1.76 [0.92 to NA] — The upper limit of CI is below the level of detection. | 5.78 [3.55 to NA] — The upper limit of CI is below the level of detection.

8. Secondary Outcome: Overall Survival (OS). Cohorts A and B, After Crossover.
Description: Overall survival (OS) is the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Time Frame: up to 3 years
Population: Participants who started on placebo and crossed over to active drug after progression.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort A: Liposarcoma Crossover; Cohort B: Osteosarcoma Crossover: Participants who started on placebo and crossed over to active drug after progression.
  Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Regorafenib: Adults: 160 mg daily; 21 days on and 7 days off Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
Arm/Group | Cohort A: Liposarcoma Crossover | Cohort B: Osteosarcoma Crossover
Number analyzed (Participants) | 15 | 11
months | 7.98 [3.98 to NA] — The upper limit of the CI is below the level of detection. | 16.11 [8.54 to NA] — The upper limit of the CI is below the level of detection.

9. Secondary Outcome: Disease Specific Survival (DSS). Cohorts A and B, After Crossover.
Description: Disease-specific survival refers to the percentage of people in a study or treatment group who have not died from a specific disease in a defined period of time.
Time Frame: up to 3 years
Population: Participants who started on placebo and crossed over to active drug upon progression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Liposarcoma Crossover | Cohort B: Osteosarcoma Crossover
Number analyzed (Participants) | 15 | 11
months | 7.98 [3.98 to NA] — The upper limit of the CI is below the level of detection. | 16.11 [8.54 to NA] — The upper limit of the CI is below the level of detection.

ADVERSE EVENTS:
Time Frame: Adverse Event data is collected beginning from the time of treatment through 30 days following cessation of treatment or until serious adverse events resolve (up to 3 years).
Description: Participants who crossed over are included in the total number at risk in the treatment arm for each Cohort as those participants were receiving treatment at time of adverse event.
Groups:
- Cohort D: Pediatric: Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
  Regorafenib
  Regorafenib:
  Pediatrics: 82mg/m2 (rounding to the nearest 20mg) daily; 21 days on and 7 days off
Arm/Group | Cohort A: Liposarcoma | Cohort A: Liposarcoma, Placebo | Cohort B: Osteosarcoma | Cohort B: Osteosarcoma, Placebo | Cohort C: Ewing Sarcoma | Cohort D: Rhabdomyosarcoma | Cohort D: Pediatric | Cohort E: Mesenchymal Chondrosarcoma
All-Cause Mortality (participants affected / at risk) | 25/39 | 7/9 | 26/33 | 8/9 | 17/30 | 4/6 | 2/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 28/39 | 7/9 | 24/33 | 7/9 | 21/30 | 4/6 | 2/4 | 0/1
Other Adverse Events (participants affected / at risk) | 26/39 | 8/9 | 26/33 | 6/9 | 22/30 | 2/6 | 1/4 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Liposarcoma (N=39) | Cohort A: Liposarcoma, Placebo (N=9) | Cohort B: Osteosarcoma (N=33) | Cohort B: Osteosarcoma, Placebo (N=9) | Cohort C: Ewing Sarcoma (N=30) | Cohort D: Rhabdomyosarcoma (N=6) | Cohort D: Pediatric (N=4) | Cohort E: Mesenchymal Chondrosarcoma (N=1)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Low Phosphate (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated AST/SGOT (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase Elevation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased WBC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hyperfibrinolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Lipase Elevation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Alkaline Phosphatase Elevated (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of Vision, Left Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Loss, Right Eye (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C/W Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colonic Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 | 0 (0)
Fatigue (General disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Failure to Thrive (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain Crisis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder Pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C. Difficile Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peri-Prosthetic Joint Infection, Left Knee (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial Thromboplastin Time Prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase Increased (Investigations) | 3 (3) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple Drug Overdose (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypophosphatemia (Investigations) | 3 (3) | 2 (2) | 5 (7) | 0 (0) | 9 (14) | 1 (1) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehyrdation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungating Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pinched nerve (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister on heel (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (2) | 3 (5) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Composite resection (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (8) | 2 (5) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Liposarcoma (N=39) | Cohort A: Liposarcoma, Placebo (N=9) | Cohort B: Osteosarcoma (N=33) | Cohort B: Osteosarcoma, Placebo (N=9) | Cohort C: Ewing Sarcoma (N=30) | Cohort D: Rhabdomyosarcoma (N=6) | Cohort D: Pediatric (N=4) | Cohort E: Mesenchymal Chondrosarcoma (N=1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 10 (19) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alkaline Phosphatase Elevated (Endocrine disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Loss, Right Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 6 (7) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 2 (2) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemina (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagesemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bloody cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 9 (11) | 0 (0) | 10 (15) | 0 (0) | 1 (1) | 0 (0)
HFS (hand and foot syndrome) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 6 (7) | 4 (9) | 5 (8) | 5 (12) | 5 (5) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT02048371/Prot_SAP_000.pdf